CLINICAL TRIAL: NCT07266155
Title: A Phase Ⅱ Extension Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of LP-005 Injection in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Efficacy, Safety, and Pharmacokinetics of LP-005 Injection in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P10-LP005-05
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP-005 1200 mg (Experimental): Patients will receive intravenous infusion of LP-005 Injection at a dose of 1200 mg once every 4 weeks.
  Interventions: Biological: LP-005 Injection
- LP-005 1500 mg (Experimental): Patients will receive intravenous infusion of LP-005 Injection at a dose of 1500 mg once every 4 weeks.
  Interventions: Biological: LP-005 Injection

INTERVENTIONS:
Biological: LP-005 Injection — IV infusion, Q4W

SUMMARY:
This is an extension study for patients who have completed a prior P10-LP005-02 clinical study. The aim of this study is to evaluate the long-term safety, efficacy, and pharmacokinetics of LP-005 injection in adult patients with paroxysmal nocturnal hemoglobinuria (PNH).

ELIGIBILITY:
Inclusion Criteria:

1. Patients have fully understood the trial, have voluntarily agreed to participate in this clinical trial, and have signed a written Informed Consent Form (ICF).
2. Patients who have completed the treatment of the Phase Ⅱ clinical study of LP-005 Injection and are assessed by the investigator as eligible for continued treatment with LP-005 Injection.
3. Patients who have received Neisseria meningitidis vaccine and Streptococcus pneumoniae vaccine in accordance with the requirements of previous studies; if the vaccine protection period does not cover the treatment duration of this study, patients must agree to receive booster vaccination in a timely manner in accordance with the vaccine administration guidelines and the requirements of local vaccination institutions.
4. Females and males of childbearing potential (including male subjects with female partners) must agree to use effective contraceptive measures from the start of the trial until 3 months after the end of the trial.

Exclusion Criteria:

1. Patients who have not completed the treatment of the Phase II clinical trial (P10-LP005-02) of the study drug.
2. Patients who have completed the Phase II treatment phase but are unwilling to continue receiving the study drug treatment.
3. Patients for whom the investigator does not recommend the continued use of LP-005 Injection after comprehensive assessment.
4. Patients who did not participate in the Phase II clinical trial (P10-LP005-02) of the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 2 years

SECONDARY OUTCOMES:
Change from baseline in serum lactate dehydrogenase (LDH) levels. | Up to approximately 2 years
Change from baseline in hemoglobin levels. | Up to approximately 2 years
Proportion of patients who are transfusion-free. | Up to approximately 2 years
Proportion of patients achieving hemoglobin levels ≥120 g/L | Up to approximately 2 years
Proportion of patients with breakthrough hemolysis | Up to approximately 2 years
Serum concentrations of LP-005. | Up to approximately 2 years
Number of patients with anti-drug antibodies (ADA) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guangsheng He, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China